CLINICAL TRIAL: NCT04300231
Title: Thoracic Epidural Analgesia Versus Rectus Sheath Block Versus Surgeon Infiltration With Liposomal Bupivacaine or Standard Bupivacaine for Post-Operative Pain Control After Cystectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Yar Yeap, Director, Acute Pain Service, Assistant Professor of Clinical Anesthesiology, Dept of Anesthesiology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1905006917
Record Dates: First submitted 2019-12-12; First posted 2020-03-09 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Cystectomy
MeSH Terms: interventions — Hydromorphone

STUDY DESIGN:
Intervention Model Description: 1. Thoracic Epidural Analgesia
  2. Rectus Sheath Block
  3. Surgeon Infiltration with Liposomal Bupivacaine
  4. Standard Bupivacaine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Thoracic epidural (Active Comparator): 1. Thoracic epidural- epidural bupivacaine 0.05%/hydromorphone 0.05mg/ml mix will be given throughout the duration of their epidural analgesia.
  Interventions: Drug: epidural bupivacaine 0.05%; Drug: /hydromorphone 0.05mg/ml
- Rectus Sheath Block (Active Comparator): 2. Rectus Sheath Block - 20 mL of Exparel® diluted with 40 mL of 0.125% bupivacaine and 40 ml of injectable saline for a total of 100 mL. The 100 mL will be injected into 4 locations below the rectus abdominis muscle.
  Interventions: Drug: Liposomal bupivacaine; Drug: bupivacaine 0.125%; Drug: injectable saline
- Surgeon Infiltration with Liposomal Bupivacaine (LB) (Active Comparator): 3. Surgeon infiltration with Liposomal Bupivacaine (LB) - 20 mL of Exparel® diluted with 40 mL of 0.125% bupivacaine and 40 ml of injectable saline for a total of 100 mL. The 100 mL will be injected throughout the incision site by the surgeon at the end of surgery, prior to abdominal wall closure.
  Interventions: Drug: Liposomal bupivacaine; Drug: bupivacaine 0.125%; Drug: injectable saline
- Surgeon Infiltration (Active Comparator): 4. Surgeon infiltration with Standard Bupivacaine (SB) - 60ml of 0.25% bupivacaine will be diluted with 40ml of saline for a total of 100ml. The 100 mL will be injected throughout the incision site by the surgeon at the end of surgery.
  Interventions: Drug: bupivacaine 0.5%; Drug: injectable saline

INTERVENTIONS:
Drug: epidural bupivacaine 0.05% — Mix of epidural bupivacaine 0.05% and hydromorphone 0.05mg/ml will be given using PCEA.
  Arms: Thoracic epidural
Drug: Liposomal bupivacaine — 20 ml
  Arms: Rectus Sheath Block; Surgeon Infiltration with Liposomal Bupivacaine (LB)
Drug: bupivacaine 0.125% — 40 mL
  Arms: Rectus Sheath Block; Surgeon Infiltration with Liposomal Bupivacaine (LB)
Drug: bupivacaine 0.5% — 60 mL
  Arms: Surgeon Infiltration
Drug: /hydromorphone 0.05mg/ml — Mix of epidural bupivacaine 0.05% and hydromorphone 0.05mg/ml will be given using PCEA.
  Arms: Thoracic epidural
Drug: injectable saline — 40 mL
  Arms: Rectus Sheath Block; Surgeon Infiltration; Surgeon Infiltration with Liposomal Bupivacaine (LB)

SUMMARY:
The purpose of this study is to compare the difference between four different pain control methods in patients who will be having a cystectomy surgery (surgical removal of the bladder).

DETAILED DESCRIPTION:
The purpose of this study is to compare the difference between four different pain control methods in patients who will be having a cystectomy surgery (surgical removal of the bladder). By collecting this data, we aim to show improved postoperative pain scores, decreased opioid needs, and decreased opioid side effects (feeling sick to your stomach, feeling drowsy/sleepy, blockage/lack of movement in the intestines, inability to completely empty the bladder, unusually slow or shallow breathing).

The specific aim of this study is to compare the difference between the pain control methods in achieving the following:

1. Decreased opioid requirements
2. Improved postoperative VAS pain scores
3. Decreased opioid side effects (Nausea, sedation, ileus, respiratory depression)
4. Decreased hospital length of stay (LOS)

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cystectomy for bladder cancer
* ASA class 1, 2, 3 or 4
* Age 18 or older, male or female
* Desires Regional anesthesia for postoperative pain control

Exclusion Criteria:

* Any contraindication for thoracic epidural.
* History of substance abuse in the past 6 months.
* Patients on more than 30mg morphine equivalents of opioids daily.
* Any physical, mental or medical conditions which in the opinion of the investigators, may confound quantifying postoperative pain resulting from surgery.
* Known allergy or other contraindications to the study medications (Acetaminophen, Gabapentin, Bupivacaine, Hydromorphone).
* Postoperative intubation.
* Any patient with history of neuropathic bowel or bladder dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2021-12-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yar Yeap, MD, Principal Investigator — Indiana University Hospital
Locations (1):
- Indiana Univeristy, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Butterworth Iv, John F., David C. Mackey, and John D. Wasnick.
- [Background] de Boer, H. D., O. Detriche, and P. Forget.
- [Background] Guo, Q., R. Li, L. Wang, D. Zhang, and Y. Ma.
- [Background] Hou, X., Z. Luo, H. Wang, Y. Zhan, L. Yang, and L. Li.
- [Background] Kalogera, E., J. N. Bakkum-Gamez, A. L. Weaver, J. P. Moriarty, B. J. Borah, C. L. Langstraat, C. J. Jankowski, et al.
- [Background] Ladjevic N, Likic-Ladjevic I, Dzamic Z, Acimovic M, Dragicevic D, Durutovic O. Combined general and epidural anaesthesia versus general anaesthesia for radical cystectomy. Acta Chir Iugosl. 2007;54(4):89-91. doi: 10.2298/aci0704089l. PMID 18595236
- [Background] Mazul-Sunko B, Gilja I, Jelisavac M, Kozul I, Troha D, Osmancevic N, El-Saleh A, Markic A, Kovacevic M, Bokarica P. Thoracic epidural analgesia for radical cystectomy improves bowel function even in traditional perioperative care: a retrospective study in eighty-five patients. Acta Clin Croat. 2014 Sep;53(3):319-25. PMID 25509242
- [Background] Ozyuvaci E, Altan A, Karadeniz T, Topsakal M, Besisik A, Yucel M. General anesthesia versus epidural and general anesthesia in radical cystectomy. Urol Int. 2005;74(1):62-7. doi: 10.1159/000082712. PMID 15711112
- [Background] ozek, J. J., M. De Ruyter, and T. W. Khan.
- [Background] Sun, J. X., K. Y. Bai, Y. F. Liu, G. Du, Z. H. Fu, H. Zhang, J. H. Yang, et al.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Thoracic Epidural | Rectus Sheath Block | Surgeon Infiltration With Liposomal Bupivacaine (LB) | Surgeon Infiltration
Started | 40 | 40 | 40 | 40
Completed | 36 | 37 | 40 | 38
Not Completed | 4 | 3 | 0 | 2
Not completed — Protocol Violation | 4 | 3 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Thoracic Epidural | Rectus Sheath Block | Surgeon Infiltration With Liposomal Bupivacaine (LB) | Surgeon Infiltration | Total
Number analyzed (Participants) | 36 | 37 | 40 | 38 | 151
Age, Continuous [Median (Full Range); unit: years] | 72 [66 to 78] | 70 [64.5 to 74] | 70 [65 to 75] | 76 [65 to 78] | 72 [64.5 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 7 | 13 | 40
  Male | 24 | 29 | 33 | 25 | 111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 36 | 37 | 40 | 38 | 151
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Body Mass Index (BMI) inkg/m^2 [Mean (Inter-Quartile Range); unit: kg/m^2] | 28.5 [24.1 to 33.7] | 27.7 [24.6 to 30.7] | 27.3 [24.7 to 29.7] | 26.8 [23.9 to 30.4] | 27.6 [24.3 to 31.1]
Duration of Surgery-in minutes [Median (Inter-Quartile Range); unit: minutes] | 305 [241 to 345] | 280.5 [246.0 to 351.0] | 285.0 [237.0 to 350.0] | 295.0 [236.0 to 357.0] | 291.4 [240 to 350.8]

OUTCOME MEASURES:

1. Primary Outcome: VAS Score at 48 Hour
Description: The VAS score will be taken with both rest and movement (knee flexion) and will be measured by a study team investigator using Visual Analog Scale (VAS). Using a scale of 0-10 for documentation with 10 being the worst pain and 0 being no pain
Time Frame: Pain scores will be measured 48 hours after surgery
Population: 48-hour Pain Scores
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Thoracic Epidural | Rectus Sheath Block | Surgeon Infiltration With Liposomal Bupivacaine (LB) | Surgeon Infiltration
Number analyzed (Participants) | 36 | 37 | 40 | 38
score on a scale
  48-hour Pain Scores at Movement | 5 [1.5 to 7.5] | 7 [4 to 8] | 4 [4 to 8] | 6 [4 to 9]
  48-hour Pain Scores at Rest | 2 [0 to 4] | 2 [1 to 5] | 3 [2 to 5] | 2 [0 to 4]

2. Primary Outcome: VAS Score at 72 Hour
Description: as for outcome 1
Time Frame: Pain scores will be measured 72 hours after surgery
Population: Pain Scores at 72 hour
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Thoracic Epidural | Rectus Sheath Block | Surgeon Infiltration With Liposomal Bupivacaine (LB) | Surgeon Infiltration
Number analyzed (Participants) | 36 | 37 | 40 | 38
score on a scale
  72-hour Pain Scores at Movement | 3.5 [1 to 5.5] | 3 [2 to 5] | 5 [4 to 7] | 4 [2 to 5]
  72-hour Pain Scores at Rest | 1 [0 to 2] | 2 [0 to 4] | 3 [1 to 6] | 2 [0 to 3]

3. Secondary Outcome: Secondary Endpoint Includes Total Opioid Consumption at 1 Hour Per PO Morphine Equivalent Dose
Description: Opioid consumption will be collected by a study team member post operatively at hour 1 per protocol time requirements
Time Frame: Opioid comsumption will be measured at 1 hour
Population: 1-hour opioid consumption
Measure: Mean (Inter-Quartile Range); unit: milligram morphine equivalents
Arm/Group | Thoracic Epidural | Rectus Sheath Block | Surgeon Infiltration With Liposomal Bupivacaine (LB) | Surgeon Infiltration
Number analyzed (Participants) | 36 | 37 | 40 | 38
milligram morphine equivalents | 5.7 [0 to 45] | 6.5 [0 to 36] | 5.8 [0 to 40] | 4.1 [0 to 42]

4. Secondary Outcome: Secondary Endpoint Includes Total Opioid Consumption at 24 Hours PO Morphine Equivalent Dose
Description: Opioid consumption will be collected by a study team member post operatively at hour 24 per protocol time requirements
Time Frame: Opioid comsumption will be measured at 24 hours
Population: Opioid consumption at 24-hour
Measure: Mean (Inter-Quartile Range); unit: milligram morphine equivalents
Arm/Group | Thoracic Epidural | Rectus Sheath Block | Surgeon Infiltration With Liposomal Bupivacaine (LB) | Surgeon Infiltration
Number analyzed (Participants) | 36 | 37 | 40 | 38
milligram morphine equivalents | 19 [12.2 to 39.1] | 36 [20 to 60] | 52 [36 to 78] | 30 [16 to 60]

5. Secondary Outcome: Secondary Endpoint Includes Total Opioid Consumption at 48 Hours PO Morphine Equivalent Dose
Description: Opioid consumption will be collected by a study team member post operatively at hour 48 per protocol time requirements
Time Frame: Opioid comsumption will be measured at 48 hours
Population: Opioid consumption at 48 hour
Measure: Mean (Inter-Quartile Range); unit: milligram morphine equivalents
Arm/Group | Thoracic Epidural | Rectus Sheath Block | Surgeon Infiltration With Liposomal Bupivacaine (LB) | Surgeon Infiltration
Number analyzed (Participants) | 36 | 37 | 40 | 38
milligram morphine equivalents | 24.8 [16.9 to 33.3] | 28 [16 to 48] | 52 [24 to 84] | 44 [20 to 96]

6. Secondary Outcome: Secondary Endpoint Includes Total Opioid Consumption at 72 Hours PO Morphine Equivalent Dose
Description: Opioid consumption will be collected by a study team member post operatively at hour 72 per protocol time requirements
Time Frame: Opioid comsumption will be measured at 72 hours
Population: Opioid consumption at 72 hour
Measure: Mean (Inter-Quartile Range); unit: milligram morphine equivalents
Arm/Group | Thoracic Epidural | Rectus Sheath Block | Surgeon Infiltration With Liposomal Bupivacaine (LB) | Surgeon Infiltration
Number analyzed (Participants) | 36 | 37 | 40 | 38
milligram morphine equivalents | 26.7 [17.8 to 36.5] | 32 [20 to 44] | 40 [24 to 72] | 32 [19 to 64]

7. Secondary Outcome: Secondary Endpoint Includes Total Opioid Consumption at 96 Hours PO Morphine Equivalent Dose
Description: Opioid consumption will be collected by a study team member post operatively at hour 96 per protocol time requirements
Time Frame: Opioid comsumption will be measured at 96 hours
Population: Opioid consumption at 96 hour
Measure: Mean (Inter-Quartile Range); unit: milligram morphine equivalents
Arm/Group | Thoracic Epidural | Rectus Sheath Block | Surgeon Infiltration With Liposomal Bupivacaine (LB) | Surgeon Infiltration
Number analyzed (Participants) | 36 | 37 | 40 | 38
milligram morphine equivalents | 21.1 [9.8 to 34.5] | 33 [15 to 55.5] | 23.3 [12 to 48] | 20 [8 to 56]

8. Secondary Outcome: VAS Score at 1 Hour
Description: as for outcome 1
Time Frame: Pain scores will be measured 1 hour after surgery
Population: 1-hour pain scores
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Thoracic Epidural | Rectus Sheath Block | Surgeon Infiltration With Liposomal Bupivacaine (LB) | Surgeon Infiltration
Number analyzed (Participants) | 36 | 37 | 40 | 38
score on a scale
  1-hour pain scores at movement | 4.4 [0 to 10] | 3.1 [0 to 10] | 2.9 [0 to 10] | 2.3 [0 to 7]
  1-hour pain scores ar rest | 3.6 [0 to 10] | 3.5 [0 to 10] | 2.7 [0 to 10] | 1.9 [0 to 7]

9. Secondary Outcome: VAS Score at 24
Description: as for outcome 1
Time Frame: Pain scores will be measured 24 hours after surgery
Population: 24-hour Pain Scores
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Thoracic Epidural | Rectus Sheath Block | Surgeon Infiltration With Liposomal Bupivacaine (LB) | Surgeon Infiltration
Number analyzed (Participants) | 36 | 37 | 40 | 38
score on a scale
  24- hour pain score at movement | 5 [1.5 to 7.5] | 7 [4 to 8] | 5 [4 to 8] | 6 [4 to 9]
  24-hour pain score at rest | 2 [0 to 5] | 3 [2 to 6] | 3 [2 to 5] | 3 [2 to 4]

10. Secondary Outcome: VAS Score at 96 Hour
Description: as for outcome 1
Time Frame: Pain scores will be measured 96 hours after surgery
Population: 96-hour pain scores
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Thoracic Epidural | Rectus Sheath Block | Surgeon Infiltration With Liposomal Bupivacaine (LB) | Surgeon Infiltration
Number analyzed (Participants) | 36 | 37 | 40 | 38
score on a scale
  96-hour pain score at movement | 4.5 [2 to 5.5] | 3 [2 to 5] | 4 [1 to 6] | 3 [1 to 4]
  96-hour pain score at rest | 2 [0 to 4] | 2 [0 to 3] | 2 [0 to 3] | 1 [0 to 3]

11. Secondary Outcome: Number of Participants With Nausea at 1 Hour
Description: Nausea scores will be collected by study team member post operatively at hour 1 per protocol. Result is reported as nausea or no nausea.
Time Frame: 1 hour
Population: 1-hour nausea score
Measure: Number; unit: participants
Arm/Group | Thoracic Epidural | Rectus Sheath Block | Surgeon Infiltration With Liposomal Bupivacaine (LB) | Surgeon Infiltration
Number analyzed (Participants) | 36 | 37 | 40 | 38
participants | 4 | 5 | 3 | 4

12. Secondary Outcome: Number of Participants With Nausea at 24 Hours
Description: Nausea scores will be collected by study team member post operatively at hour 24 per protocol. Result is reported as nausea or no nausea.
Time Frame: 24 hour
Population: 24-hour nausea score
Measure: Number; unit: participants
Arm/Group | Thoracic Epidural | Rectus Sheath Block | Surgeon Infiltration With Liposomal Bupivacaine (LB) | Surgeon Infiltration
Number analyzed (Participants) | 36 | 37 | 40 | 38
participants | 9 | 5 | 7 | 9

13. Secondary Outcome: Number of Participants With Nausea at 48 Hours
Description: Nausea scores will be collected by study team member post operatively at hour 48 per protocol. Result is reported as nausea or no nausea.
Time Frame: 48 hour
Population: 48-hour nausea score
Measure: Number; unit: participants
Arm/Group | Thoracic Epidural | Rectus Sheath Block | Surgeon Infiltration With Liposomal Bupivacaine (LB) | Surgeon Infiltration
Number analyzed (Participants) | 36 | 37 | 40 | 38
participants | 11 | 11 | 10 | 13

14. Secondary Outcome: Number of Participants With Nausea at 72 Hours
Description: Nausea scores will be collected by study team member post operatively at hour 72 per protocol. Result is reported as nausea or no nausea.
Time Frame: 72 hour
Population: 72-hour nausea score
Measure: Number; unit: participants
Arm/Group | Thoracic Epidural | Rectus Sheath Block | Surgeon Infiltration With Liposomal Bupivacaine (LB) | Surgeon Infiltration
Number analyzed (Participants) | 36 | 37 | 40 | 38
participants | 11 | 12 | 17 | 18

15. Secondary Outcome: Number of Participants With Nausea at 96 Hours
Description: Nausea scores will be collected by study team member post operatively at hour 96 per protocol. Result is reported as nausea or no nausea.
Time Frame: 96 hour
Population: 96-hour nausea score
Measure: Number; unit: participants
Arm/Group | Thoracic Epidural | Rectus Sheath Block | Surgeon Infiltration With Liposomal Bupivacaine (LB) | Surgeon Infiltration
Number analyzed (Participants) | 36 | 37 | 40 | 38
participants | 15 | 6 | 12 | 14

16. Secondary Outcome: Number of Participants With Sedation at 1 Hour
Description: Sedation scores will be collected by a study team member post operatively at hour 1. Results are interpreted as patient with or without any sedation.
Time Frame: 1 hour
Population: 1hr sedation score
Measure: Number; unit: participants
Arm/Group | Thoracic Epidural | Rectus Sheath Block | Surgeon Infiltration With Liposomal Bupivacaine (LB) | Surgeon Infiltration
Number analyzed (Participants) | 36 | 37 | 40 | 38
participants | 2 | 2 | 2 | 2

17. Secondary Outcome: Number of Participants With Sedation at 24 Hours
Description: Sedation scores will be collected by a study team member post operatively at hour 24. Results are interpreted as patient with or without any sedation.
Time Frame: 24 hour
Population: 24-hour sedation score
Measure: Number; unit: participants
Arm/Group | Thoracic Epidural | Rectus Sheath Block | Surgeon Infiltration With Liposomal Bupivacaine (LB) | Surgeon Infiltration
Number analyzed (Participants) | 36 | 37 | 40 | 38
participants | 1 | 0 | 0 | 0

18. Secondary Outcome: Number of Participants With Sedation at 48 Hours
Description: Sedation scores will be collected by a study team member post operatively at hour 48. Results are interpreted as patient with or without any sedation.
Time Frame: 48 hour
Population: 48-hour sedation score
Measure: Number; unit: participants
Arm/Group | Thoracic Epidural | Rectus Sheath Block | Surgeon Infiltration With Liposomal Bupivacaine (LB) | Surgeon Infiltration
Number analyzed (Participants) | 36 | 37 | 40 | 38
participants | 2 | 1 | 2 | 0

19. Secondary Outcome: Number of Participants With Sedation at 72 Hours
Description: Sedation scores will be collected by a study team member post operatively at hour 72. Results are interpreted as patient with or without any sedation.
Time Frame: 72 hour
Population: 72-hour sedation score
Measure: Number; unit: participants
Arm/Group | Thoracic Epidural | Rectus Sheath Block | Surgeon Infiltration With Liposomal Bupivacaine (LB) | Surgeon Infiltration
Number analyzed (Participants) | 36 | 37 | 40 | 38
participants | 0 | 1 | 2 | 1

20. Secondary Outcome: Number of Participants With Sedation at 96 Hours
Description: Sedation scores will be collected by a study team member post operatively at hour 96. Results are interpreted as patient with or without any sedation.
Time Frame: 96 hour
Population: 96-hour sedation score
Measure: Number; unit: participants
Arm/Group | Thoracic Epidural | Rectus Sheath Block | Surgeon Infiltration With Liposomal Bupivacaine (LB) | Surgeon Infiltration
Number analyzed (Participants) | 36 | 37 | 40 | 38
participants | 1 | 1 | 0 | 2

21. Secondary Outcome: First Flatus-bowel Movement
Description: The first time the patients passes gas post operatively.
Time Frame: Assess daily until patient passes gas postoperatively, up to 120 hours after surgery
Population: Time to first Flatus
Measure: Mean (Inter-Quartile Range); unit: Hours
Arm/Group | Thoracic Epidural | Rectus Sheath Block | Surgeon Infiltration With Liposomal Bupivacaine (LB) | Surgeon Infiltration
Number analyzed (Participants) | 36 | 37 | 40 | 38
Hours | 70.3 [42.8 to 89.6] | 55.5 [34.5 to 84] | 69.7 [56.2 to 96.7] | 59.8 [37.7 to 78.4]

22. Secondary Outcome: Postoperative Creatinine
Description: Lab level of Creatinine will be recorded for 4 days post operatively.
Time Frame: Creatinine level will be collected daily postoperatively for 4 days
Population: creatinine level Postoperatively
Measure: Mean (Inter-Quartile Range); unit: mg/dL
Arm/Group | Thoracic Epidural | Rectus Sheath Block | Surgeon Infiltration With Liposomal Bupivacaine (LB) | Surgeon Infiltration
Number analyzed (Participants) | 36 | 37 | 40 | 38
mg/dL | 1.0 [0.80 to 1.38] | 0.98 [0.79 to 1.25] | 1.08 [0.79 to 1.46] | 0.96 [0.78 to 1.28]

23. Secondary Outcome: Time to Discharge-Length of Stay
Description: Length of Stay will be collected from Cerner Electronic Medical Record. Pt. followed for length of stay, up till 4 weeks after surgery.
Time Frame: From hospital admission to discharge time
Population: Length of Stay (LOS)
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | Thoracic Epidural | Rectus Sheath Block | Surgeon Infiltration With Liposomal Bupivacaine (LB) | Surgeon Infiltration
Number analyzed (Participants) | 36 | 37 | 40 | 38
days | 7.1 [6.1 to 8.9] | 6.0 [5.1 to 7.1] | 6.4 [5.3 to 8.2] | 7.0 [6.1 to 9.1]

24. Secondary Outcome: Incidence of Hypotension
Description: Defined as BP decrease of more than 20% from baseline. The reported number for each arm is the cumulative number of hypotension episodes experienced in each arm.
Time Frame: number of times hypotension occurred the first 96 hours after surgery.
Population: cumulative number of hypotension episodes in 96 hours
Measure: Number; unit: hypotension episodes
Arm/Group | Thoracic Epidural | Rectus Sheath Block | Surgeon Infiltration With Liposomal Bupivacaine (LB) | Surgeon Infiltration
Number analyzed (Participants) | 36 | 37 | 40 | 38
hypotension episodes | 25 | 22 | 16 | 26

25. Secondary Outcome: Incidence of Respiratory Depression
Description: Define by use of Narcan
Time Frame: assess daily as yes/no up to 96hr
Population: Incidence of Respiratory Depression
Measure: Count of Participants; unit: Participants
Arm/Group | Thoracic Epidural | Rectus Sheath Block | Surgeon Infiltration With Liposomal Bupivacaine (LB) | Surgeon Infiltration
Number analyzed (Participants) | 36 | 37 | 40 | 38
Participants | 0 | 1 | 2 | 1

26. Secondary Outcome: Ambulation Activity Postoperatively
Description: Number of participants who got out of bed and is ambulatory on Postoperative Day 1 and postoperative Day 2
Time Frame: Patients followed for ambulation activities on postop Day 1 and Day 2
Population: Ambulation activity
Measure: Count of Participants; unit: Participants
Arm/Group | Thoracic Epidural | Rectus Sheath Block | Surgeon Infiltration With Liposomal Bupivacaine (LB) | Surgeon Infiltration
Number analyzed (Participants) | 36 | 37 | 40 | 38
Participants
  Patient Starts ambulating on Day 1-Yes | 34 | 35 | 38 | 36
  Patient starts ambulating on Day 2-yes | 1 | 1 | 2 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected for up to 3 weeks of hospitalization stay
Arm/Group | Thoracic Epidural | Rectus Sheath Block | Surgeon Infiltration With Liposomal Bupivacaine (LB) | Surgeon Infiltration
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 4/40 | 8/40 | 2/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thoracic Epidural (N=40) | Rectus Sheath Block (N=40) | Surgeon Infiltration With Liposomal Bupivacaine (LB) (N=40) | Surgeon Infiltration (N=40)
Ileus (Gastrointestinal disorders) | 0 (0) | 2 (4) | 7 (8) | 2 (2)
respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) — defined as narcan used for respiratory depression

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-21): https://cdn.clinicaltrials.gov/large-docs/31/NCT04300231/Prot_SAP_002.pdf